CLINICAL TRIAL: NCT05818124
Title: A Phase 2a Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of MK-4482 in Healthy Participants Inoculated With Experimental Influenza Virus
Brief Title: Efficacy and Safety of Molnupiravir in Healthy Participants Inoculated With Experimental Influenza Virus (MK-4482-019)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4482-019
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Influenza Infection
MeSH Terms: interventions — molnupiravir; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Panel A: Molnupiravir Post-Exposure Prophylaxis (Part 2) (Experimental): Molnupiravir 800 mg every 12 hours Day 0 PM through Day 5 AM, placebo molnupiravir every 12 hours Day 5 PM through Day 6 PM
  Interventions: Drug: Molnupiravir; Drug: Placebo molnupiravir; Biological: Influenza A Virus
- Panel B: Molnupiravir Treatment (Part 2) (Experimental): Placebo molnupiravir every 12 hours Day 0 PM through Day 1 PM, molnupiravir 800 mg every 12 hours Day 2 AM through Day 6 PM
  Interventions: Drug: Molnupiravir; Drug: Placebo molnupiravir; Biological: Influenza A Virus
- Panel C: Oseltamivir Treatment (Part 2) (Active Comparator): Placebo oseltamivir Day 0 PM through Day 1 PM, oseltamivir 75 mg plus placebo so the total number of capsules is always 4 per dose every 12 hours Day 2 AM through Day 6 PM
  Interventions: Drug: Placebo oseltamivir; Drug: Oseltamivir; Biological: Influenza A Virus
- Panel D: Molnupiravir Placebo (Part 2) (Placebo Comparator): Placebo molnupiravir every 12 hours Day 0 PM through Day 6 PM
  Interventions: Drug: Placebo molnupiravir; Biological: Influenza A Virus
- Virus Inoculation (Part 1 & 2) (Experimental): Influenza A challenge virus given once by intranasal administration
  Interventions: Biological: Influenza A Virus

INTERVENTIONS:
Drug: Molnupiravir — Four molnupiravir 200 mg capsules (800 mg total dose) taken twice daily by mouth.
  Other Names: MK-4482
  Arms: Panel A: Molnupiravir Post-Exposure Prophylaxis (Part 2); Panel B: Molnupiravir Treatment (Part 2)
Drug: Placebo molnupiravir — Four placebo capsules matched to molnupiravir taken twice daily by mouth.
  Arms: Panel A: Molnupiravir Post-Exposure Prophylaxis (Part 2); Panel B: Molnupiravir Treatment (Part 2); Panel D: Molnupiravir Placebo (Part 2)
Drug: Placebo oseltamivir — Placebo capsule matched to oseltamivir taken twice daily by mouth.
  Arms: Panel C: Oseltamivir Treatment (Part 2)
Drug: Oseltamivir — One capsule of oseltamivir 75 mg taken twice daily by mouth.
  Arms: Panel C: Oseltamivir Treatment (Part 2)
Biological: Influenza A Virus — Influenza A challenge virus given once by intranasal administration at an inoculum concentration of between approximately 5 and 7 Log10 tissue culture infective dose 50% (TCID50/mL).

SUMMARY:
This is a phase 2a double-blind, randomized, placebo-controlled study to evaluate the efficacy and safety of molnupiravir (MK-4482) in healthy participants inoculated with experimental influenza virus. The primary hypotheses are that MK-4482 initiated 12 hours following intranasal inoculation of the influenza challenge virus reduces the peak viral load compared to placebo and that MK-4482 initiated 2 days following intranasal inoculation of the influenza challenge virus reduces the viral load area under the curve (AUC) compared to placebo.

DETAILED DESCRIPTION:
This study has two parts. Part 1 is an open-label validation study, with a cohort of 20 untreated participants undergoing nasal inoculation with the A/France/759/21 [H1N1] strain on Day 0 to confirm viral infectivity and disease. Part 2 will be a randomized, double-blind placebo- and active-comparator-controlled study where participants will be inoculated on Day 0 with either the A/France/759/21 [H1N1] virus used in Part 1 or an alternative influenza virus. Part 2 will evaluate the antiviral efficacy, pharmacokinetics, and safety of MK-4482 in participants inoculated with the challenge virus.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health based on medical history, physical examination, vital sign measurements, spirometry, and electrocardiograms performed before inoculation.
* Has a total body weight ≥50 kg and Body Mass Index (BMI) ≥18 kg/m^2 and ≤35 kg/m^2.
* For males: abstains from heterosexual intercourse as their preferred and usual lifestyle and agrees to remain abstinent OR uses contraception unless confirmed to be azoospermic.
* For participants assigned female sex at birth: is not pregnant or breastfeeding, AND is either not a person of childbearing potential (POCBP) or is a POCBP AND uses a contraceptive method that is highly effective (low user dependency method, OR a user dependent hormonal method in combination with barrier method), or is abstinent from penile-vaginal intercourse as their preferred and usual lifestyle, has a negative highly sensitive pregnancy test, abstains from breastfeeding, and has medical, menstrual, and recent sexual activity history reviewed by the investigator to decrease risk of early undetected pregnancy.

Exclusion Criteria:

* Has a history of, or has currently active, symptoms or signs suggestive of upper or lower respiratory tract infection within 4 weeks prior to admission to quarantine.
* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological abnormalities or diseases.
* Is mentally or legally incapacitated, has significant emotional problems at the time of prestudy visit, or expected during the conduct of the study, or has a history of clinically significant psychiatric disorder of the last 5 years.
* Has a history of cancer.
* Has a history of rhinitis which is clinically active, or history of moderate to severe rhinitis, or history of seasonal allergic rhinitis likely to be active at the time of inclusion into the study and/or requiring regular nasal corticosteroids on an at least weekly basis, within 30 days prior to admission to quarantine.
* Has a history of atopic dermatitis/eczema which is clinically severe and/or requiring moderate to large amounts of daily dermal corticosteroids.
* Has a diagnosis of cluster headache/migraine or is receiving prophylaxis against migraine.
* Has a lifetime history of anaphylaxis and/or a lifetime history of severe allergic reaction. Significant intolerance to any food or drug in the last 12 months.
* Has had major surgery and/or donated or lost 1 unit of blood within 3 months prior to the prestudy visit.
* Uses or anticipates the use of concomitant medications, including vitamins or herbal and dietary supplements from approximately 2 weeks prior to the planned date of viral challenge until the poststudy visit.
* Has evidence of receipt of vaccine within the 4 weeks prior to the planned date of viral challenge.
* Intends to receive any vaccine(s) before the last day of follow-up.
* Has received any investigational drug within 3 months prior to the planned date of viral challenge.
* Has received 3 or more investigational drugs within the previous 12 months prior to the planned date of viral challenge.
* Has had prior inoculation with a virus from the same virus subtype as the challenge virus.
* Has had prior inoculation with a virus from the same virus-family as the challenge virus in the last 12 months.
* Has had prior participation in another human viral challenge study with a respiratory virus in the preceding 3 months, taken from the date of viral challenge in the previous study to the date of expected viral challenge in this study.
* Has smoked ≥10 pack-years at any time.
* Has a recent history or presence of alcohol addiction, or excessive use of alcohol.
* Consumes excessive amounts, defined as more than 6 servings of caffeinated beverages or xanthine-containing products.
* Has any significant abnormality altering the anatomy of the nose in a substantial way or nasopharynx that may interfere with the aims of the study and, in particular, any of the nasal assessments or viral challenge.
* Has any clinically significant history of epistaxis.
* Has had any nasal or sinus surgery within 3 months.
* Is a regular user of cannabis or any illicit drugs, or has a history of drug abuse within approximately 1 year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- hVIVO Services ( Site 0001), London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-part study in healthy participants. Part 1 was an open label validation study to confirm that Part 2 can proceed using the same challenge strain.
Pre-assignment Details: Before viral inoculation on Day 0, participants had serosuitability confirmed by negative hemagglutination inhibition and quarantined participants underwent additional screening to exclude those with respiratory pathogens, and participants who were excluded at this time did not receive study intervention.
Groups:
- Viral Inoculation (Part 1): Participants were nasally inoculated with a single inoculum titer of 10^6.26 TCID50 (tissue culture infective dose (50%))/mL of A/France/759/21 [H1N1] strain on Day 0 to confirm viral infectivity and disease.
- Molnupiravir Post-Exposure Prophylaxis (PEP): Participants received 800 mg molnupiravir orally every 12 hours (Q12H) for 5 days beginning on Day 0 PM (~12 h after inoculation with A/France/759/21 [H1N1] virus). Participants switched to oral placebo beginning on Day 5 PM to Day 6 PM.
- Molnupiravir Treatment (Tx): Participants received placebo Q12H beginning on Day 0 PM through Day 1 PM. Participants switched to 800 mg Molnupiravir beginning on Day 2 AM (~ 2 days after inoculation with A/France/759/21 [H1N1] virus) to Day 6 PM.
- Oseltamivir (OTV) Tx: Participants received placebo Q12H orally beginning on Day 0 PM through Day 1 PM. Participants switched to 75 mg OTV orally beginning on Day 2 AM (~ 2 days after inoculation with A/France/759/21 [H1N1] virus) to Day 6 PM.
- Placebo: Participants received placebo Q12H orally beginning from Day 0 PM through Day 6 PM.
Period: Part 1: Validation
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Started | 20 | 0 | 0 | 0 | 0
Completed | 20 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Started | 0 (Part 1 enrollment was strictly for characterization of the viral strain and participants did not receive study drug nor enroll in period 2.) | 35 (Part 2 enrollment consisted of a different cohort than Part 1 using the challenge virus from Part 1 to evaluate performance of MK-4482 in the challenge model.) | 36 (Part 2 enrollment consisted of a different cohort than Part 1 using the challenge virus from Part 1 to evaluate performance of MK-4482 in the challenge model.) | 35 (Part 2 enrollment consisted of a different cohort than Part 1 using the challenge virus from Part 1 to evaluate performance of MK-4482 in the challenge model.) | 35 (Part 2 enrollment consisted of a different cohort than Part 1 using the challenge virus from Part 1 to evaluate performance of MK-4482 in the challenge model.)
Completed | 0 | 35 | 36 | 35 | 35
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Oseltamivir (OTV) Tx: Participants received placebo Q12H beginning on Day 0 PM through Day 1 PM. Participants switched to 75 mg OTV beginning on Day 2 AM (~ 2 days after inoculation with A/France/759/21 [H1N1] virus) to Day 6 PM.
- Placebo: Participants received placebo Q12H beginning from Day 0 PM through Day 6 PM
- Total: Total of all reporting groups
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo | Total
Number analyzed (Participants) | 20 | 35 | 36 | 35 | 35 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 35 | 36 | 35 | 35 | 161
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.8 (9.5) | 28.6 (6.8) | 29.3 (8.3) | 31.5 (9.2) | 30.8 (8.5) | 30.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 17 | 12 | 18 | 71
  Male | 11 | 20 | 19 | 23 | 17 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 2 | 1 | 9
  Not Hispanic or Latino | 18 | 33 | 33 | 33 | 34 | 151
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 1 | 2 | 4 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 2 | 1 | 3 | 12
  White | 13 | 28 | 32 | 28 | 24 | 125
  More than one race | 2 | 0 | 1 | 4 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Part 1: QVC-Confirmed Influenza Infection From Day 1 PM Through Day 8 AM After Intranasal Inoculation
Description: QVC-Confirmed Influenza Infection was defined as the number of participants with one quantifiable ≥LLOQ influenza challenge virus measurement from QVC (plaque assay) of nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening). QVC confirmed influenza infection in Part 1 participants from day 1 PM up to day 8 post viral inoculation is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
Participants | 15 |  |  |  |

2. Secondary Outcome: Part 1: QVC-Confirmed Influenza Infection From Day 2 PM Through Day 8 AM After Intranasal Inoculation
Description: QVC-Confirmed Influenza Infection was defined as the number of participants with one quantifiable ≥LLOQ influenza challenge virus measurement from QVC (plaque assay) of nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening). QVC confirmed influenza infection in Part 1 participants from day 2 PM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 2 PM Up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
Participants | 8 |  |  |  |

3. Secondary Outcome: Part 1: VL-AUC Determined by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation
Description: VL-AUC is the area under the viral load-time curve of influenza challenge virus nasopharyngeal samples determined by qRT-PCR. H1N1 viral load was computed for each participant from nasopharyngeal samples collected twice daily (morning and evening) from day 1 PM to day 8 AM. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: Day 1 PM, Days 2, 3, 4, 5, 6, 7 - twice daily (AM and PM), and day 8 AM post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (95% Confidence Interval); unit: day*log10 copies/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
day*log10 copies/mL | 17.29 [13.57 to 21.01] |  |  |  |

4. Secondary Outcome: Part 1: VL-AUC Determined by qRT-PCR From Day 2 PM Through Day 8 AM After Intranasal Inoculation
Description: VL-AUC is the area under the viral load-time curve of influenza challenge virus nasopharyngeal samples determined by qRT-PCR. H1N1 viral load was computed for each participant from nasopharyngeal samples collected twice daily (morning and evening) from day 2 PM to day 8 AM. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for part 1 participants were presented for this endpoint. VL-AUC by qRT-PCR in Part 1 participants from day 2 PM up to day 8 is presented.
Time Frame: Day 2 PM, Days 3, 4, 5, 6, 7 - twice daily (AM and PM), and day 8 AM post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (95% Confidence Interval); unit: day*log10 copies/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
day*log10 copies/mL | 12.29 [9.41 to 15.18] |  |  |  |

5. Secondary Outcome: Part 1: VL-AUC Determined by Quantitative Viral Culture (TCID50 Assay) From Day 1 PM Through Day 8 AM After Intranasal Inoculation
Description: VL-AUC is the area under the viral load-time curve of influenza challenge virus nasopharyngeal samples determined by QVC. H1N1 viral load was computed for each participant from nasophayngeal samples collected twice daily (morning and evening) from day 1 PM to day 8 AM. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for part 1 participants were presented for this endpoint. VL-AUC by QVC in Part 1 participants from day 1 PM up to day 8 is presented.
Time Frame: Day 1 PM, Days 2, 3, 4, 5, 6, 7 - twice daily (AM and PM), and day 8 AM post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (95% Confidence Interval); unit: day*log10 TCID 50/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
day*log10 TCID 50/mL | 5.45 [3.88 to 7.01] |  |  |  |

6. Secondary Outcome: Part 1: VL-AUC Determined by Quantitative Viral Culture (TCID50 Assay) From Day 2 PM Through Day 8 AM After Intranasal Inoculation
Description: VL-AUC is the area under the viral load-time curve of influenza challenge virus nasopharyngeal samples determined by QVC. H1N1 viral load was computed for each participant from nasopharyngeal samples collected twice daily (morning and evening) from day 1 PM to day 8 AM. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for part 1 participants were presented for this endpoint. VL-AUC by QVC in Part 1 participants from day 2 PM up to day 8 is presented.
Time Frame: Day 2 PM, Days 3, 4, 5, 6, 7 - twice daily (AM and PM), and day 8 AM post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (95% Confidence Interval); unit: day*log10 copies/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
day*log10 copies/mL | 2.27 [1.28 to 3.26] |  |  |  |

7. Secondary Outcome: Part 1: PVL Determined by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation
Description: PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening) from day 1 PM (baseline) through day 8 AM. PVL of the H1N1 strain was measured by qRT-PCR and analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
log10 copies/mL | 5.89 [4.89 to 6.88] |  |  |  |

8. Secondary Outcome: Part 1: PVL Determined by qRT-PCR From Day 2 PM Through Day 8 AM After Intranasal Inoculation
Description: PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening) from day 2 PM (baseline) through day 8 AM. PVL of the H1N1 strain was measured by qRT-PCR and analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 2 PM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
log10 copies/mL | 5.15 [4.31 to 5.99] |  |  |  |

9. Secondary Outcome: Part 1: PVL Determined by Quantitative Viral Culture (TCID50 Assay) From Day 1 PM Through Day 8 AM After Intranasal Inoculation
Description: PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening) from day 1 PM (baseline) through day 8 AM. PVL of the H1N1 strain was measured by QVC and analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (95% Confidence Interval); unit: log10 TCID 50/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
log10 TCID 50/mL | 4.05 [3.30 to 4.81] |  |  |  |

10. Secondary Outcome: Part 1: PVL Determined by Quantitative Viral Culture (TCID50 Assay) From Day 2 PM Through Day 8 AM After Intranasal Inoculation
Description: PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening) from day 2 PM (baseline) through day 8 AM. PVL of the H1N1 strain was measured by QVC and analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 2 PM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (95% Confidence Interval); unit: log10 TCID 50/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
log10 TCID 50/mL | 2.33 [1.54 to 3.13] |  |  |  |

11. Secondary Outcome: Part 1: Duration in Days of Quantifiable Influenza Infection by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation
Description: Duration in days of quantifiable influenza infection was defined as the time in days from the first quantifiable (≥LLOQ) influenza challenge virus measurement until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure (after which there are no more confirmed quantifiable samples) determined by qRT-PCR from nasal wash samples collected twice daily (morning and evening). Duration of Quantifiable Influenza by qRT-PCR in Part 1 participants from day 1 PM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 15 | 0 | 0 | 0 | 0
Days | 3.23 (1.42) |  |  |  |

12. Secondary Outcome: Part 1: Duration in Days of Quantifiable Influenza Infection by qRT-PCR From Day 2 PM Through Day 8 AM After Intranasal Inoculation
Description: Duration in days of quantifiable influenza infection was defined as the time in days from the first quantifiable (≥LLOQ) influenza challenge virus measurement until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure after which there are no more confirmed quantifiable samples) determined by qRT-PCR from nasal wash samples collected twice daily (morning and evening). Duration of Quantifiable Influenza by qRT-PCR in Part 1 participants from day 2 PM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 2 PM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 14 | 0 | 0 | 0 | 0
Days | 2.24 (1.52) |  |  |  |

13. Secondary Outcome: Part 1: Duration in Days of Quantifiable Influenza Infection by QVC (TCID50 Assay) Confirmed Infection From Day 1 PM Through Day 8 AM After Intranasal Inoculation
Description: Duration in days of quantifiable influenza infection was defined as the time in days from the first quantifiable (≥LLOQ) influenza challenge virus measurement until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure after which there are no more confirmed quantifiable samples) determined by QVC (plaque assay) from nasal wash samples collected twice daily (morning and evening). Duration of Quantifiable Influenza by QVC in Part 1 participants from day 1 PM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 15 | 0 | 0 | 0 | 0
Days | 1.10 (1.01) |  |  |  |

14. Secondary Outcome: Part 1: Duration in Days of Quantifiable Influenza Infection by QVC Confirmed Infection From Day 2 PM Through Day 8 AM After Intranasal Inoculation
Description: Duration in days of quantifiable influenza infection was defined as the time in days from the first quantifiable (≥LLOQ) influenza challenge virus measurement until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure after which there are no more confirmed quantifiable samples) determined by QVC (plaque assay) from nasal wash samples collected twice daily (morning and evening). Duration of Quantifiable Influenza by QVC in Part 1 participants from day 2 PM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 2 PM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
Days | 0.79 (1.11) |  |  |  |

15. Secondary Outcome: Part 1: Area Under the Total Symptom Score-Time Curve (TSS-AUC) From Day 1 AM Through Day 8 AM After Intranasal Inoculation
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom was used to obtain a total symptom score (TSS). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. TSS were used to calculate the AUC for each participant based on the available non-missing calculated total symptom scores between Day 1 until Day 8 (quarantine discharge) using the Trapezoidal rule. TSS-AUC measured from 10 symptoms assessed 3 times daily within the graded symptom scoring was reported. TSS-AUC in Part 1 participants from day 1 AM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 1 AM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (95% Confidence Interval); unit: Scores on a Scale*Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
Scores on a Scale*Days | 23.48 [14.89 to 32.08] |  |  |  |

16. Secondary Outcome: Part 1: Area Under the Total Symptom Score-Time Curve (TSS-AUC) From Day 2 AM Through Day 8 AM After Intranasal Inoculation
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom was used to obtain TSS. Total symptom scores (TSS) ranged from 0 to 31, with higher scores indicating greater symptom severity. TSS were used to calculate the AUC for each participant based on the available non-missing calculated total symptom scores between Day 2 until Day 8 (quarantine discharge) using the Trapezoidal rule. TSS-AUC in Part 1 participants from day 2 AM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (95% Confidence Interval); unit: Scores on a Scale*Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
Scores on a Scale*Days | 16.95 [9.62 to 24.28] |  |  |  |

17. Secondary Outcome: Part 1: Peak Total Symptom Score (TSS) From Day 1 AM Through Day 8 AM After Intranasal Inoculation
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom was used to obtain a total symptom score (TSS). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. The highest TSS (defined as the sum of all 10 individual composite symptoms) was summarized by treatment group and analyzed using a linear model with treatment group as a fixed categorical effect. Peak TSS measured from 10 symptoms within the graded symptom scoring system collected 3 times daily was reported. Peak TSS in Part 1 participants from day 1 AM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 1 AM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
Scores on a Scale | 9.65 [6.94 to 12.36] |  |  |  |

18. Secondary Outcome: Part 1: Peak Total Symptom Score (TSS) From Day 2 AM Through Day 8 AM After Intranasal Inoculation
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom was used to obtain TSS. TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. The highest TSS (defined as the sum of all 10 individual composite symptoms) was summarized by treatment group and analyzed using a linear model with treatment group as a fixed categorical effect. Peak TSS measured from 10 symptoms within the graded symptom scoring system collected 3 times daily was reported. Peak TSS in Part 1 participants from day 2 AM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
Scores on a Scale | 8.85 [6.03 to 11.67] |  |  |  |

19. Secondary Outcome: Part 1: Daily Maximum TSS From Day 1 AM Through Day 8 AM After Intranasal Inoculation
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom was used to obtain TSS. TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. Maximum TSS on each day, measured by graded symptom scoring system collected 3 times daily were reported. Daily maximum TSS in Part 1 participants from day 1 AM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 1 AM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
Scores on a Scale
  Day 1 | 6.15 (4.23) |  |  |  |
  Day 2 | 8.65 (4.91) |  |  |  |
  Day 3 | 6.80 (5.61) |  |  |  |
  Day 4 | 4.85 (5.49) |  |  |  |
  Day 5 | 2.90 (3.74) |  |  |  |
  Day 6 | 2.05 (2.52) |  |  |  |
  Day 7 | 0.70 (1.45) |  |  |  |
  Day 8 | 0.45 (1.47) |  |  |  |

20. Secondary Outcome: Part 1: Duration in Days of Grade ≥2 Symptoms From Day 1 AM Through Day 8 AM After Intranasal Inoculation
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from Grade 0 ("no symptoms") to Grade 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from Grade 0 ("no symptoms") to Grade 4 ("symptoms at rest"). Duration of Grade 2 symptoms is defined as the duration in days from the first occurrence of a Grade 2 or higher symptom until the first 24 hours period where no Grade 2 or higher symptoms are recorded. Duration in days of grade ≥2 Symptoms in part 1 participants from day 1 AM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 1 AM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 14 | 0 | 0 | 0 | 0
Days | 2.65 (1.38) |  |  |  |

21. Secondary Outcome: Part 1: Duration of Grade ≥2 Symptoms From Day 2 AM Through Day 8 AM After Intranasal Inoculation
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from Grade 0 ("no symptoms") to Grade 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from Grade 0 ("no symptoms") to Grade 4 ("symptoms at rest"). Duration of Grade 2 symptoms is defined as the duration in days from the first occurrence of a Grade 2 or higher symptom until the first 24 hours period where no Grade 2 or higher symptoms are recorded. Duration in days of grade ≥2 Symptoms in part 1 participants from day 2 AM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 14 | 0 | 0 | 0 | 0
Days | 1.84 (1.35) |  |  |  |

22. Secondary Outcome: Part 1: Time to Symptom Resolution From Day 1 AM Through Day 8 AM After Intranasal Inoculation
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. Time in days to symptom resolution was defined as the time in days from the beginning of the specified time frame until the beginning of a 24-hour period with no symptoms above the baseline maximum TSS, as measured by graded symptom scoring system collected 3 times daily. Baseline maximum is defined as the maximum TSS on Day -1 (1 day prior to intranasal inoculation). Time in days to symptom resolution in part 1 participants from day 1 AM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 1 AM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
Days | 4.15 (2.44) |  |  |  |

23. Secondary Outcome: Part 1: Time to Symptom Resolution From Day 2 AM Through Discharge From Quarantine (Day 8 AM) After Intranasal Inoculation
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. Time in days to symptom resolution was defined as the time (in days) from the beginning of the specified time frame until the beginning of a 24-hour period with no symptoms above the baseline maximum TSS, as measured by graded symptom scoring system collected 3 times daily. Baseline maximum is defined as the maximum TSS on Day -1 (1 day prior to intranasal inoculation). Time in days to symptom resolution in part 1 participants from day 2 AM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
Days | 3.21 (2.03) |  |  |  |

24. Secondary Outcome: Part 1: Time to Peak TSS From Day 1 AM Through Day 8 AM After Intranasal Inoculation
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom was used to obtain TSS. TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. The highest total symptom score recorded on each day, across the three assessments, for each participant was summarized descriptively by treatment group and assessment day. Time to peak TSS was defined as the time from the assessment at Day 1 AM until the highest total symptom score was calculated. Time to peak TSS in Part 1 participants from day 1 AM up to day 8 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 1 AM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 19 | 0 | 0 | 0 | 0
Days | 1.24 (0.76) |  |  |  |

25. Secondary Outcome: Part 2: VL-AUC Determined by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: VL-AUC is the area under the viral load-time curve of influenza challenge virus nasopharyngeal samples determined by qRT-PCR. H1N1 viral load was computed for each participant from nasopharyngeal samples collected twice daily (morning and evening) from day 1 PM to day 8 AM. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: Day 1 PM, Days 2, 3, 4, 5, 6, 7 - twice daily (AM and PM), and day 8 AM post viral inoculation
Population: All randomized participants who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation and had available data for the endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: day*log10 copies/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
day*log10 copies/mL |  | 11.10 [8.64 to 13.57] |  |  | 11.58 [9.12 to 14.05]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other; p = 0.783, ANOVA; Difference in Least Squares Mean = -0.48, 95% CI 2-sided [-3.97 to 3.00]

26. Secondary Outcome: Part 2: VL-AUC Determined by Quantitative Viral Culture (TCID50 Assay) From Day 1 PM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: VL-AUC is the area under the viral load-time curve of influenza challenge virus nasopharyngeal samples determined by QVC. H1N1 viral load was computed for each participant from nasophayngeal samples collected twice daily (morning and evening) from day 1 PM to day 8 AM. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: Day 1 PM, Days 2, 3, 4, 5, 6, 7 - twice daily (AM and PM), and day 8 AM post viral inoculation
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: day*log10 TCID50/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 17 | 0 | 0 | 16
day*log10 TCID50/mL |  | 2.15 [0.76 to 3.54] |  |  | 4.36 [2.92 to 5.79]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other; p = 0.032, ANOVA; Difference in Least Squares Mean = -2.21, 95% CI 2-sided [-4.21 to -0.21]

27. Secondary Outcome: Part 2: PVL Determined by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening) from day 1 PM (baseline) through day 8 AM. PVL of the H1N1 strain was measured by qRT-PCR and analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: All randomized participants who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into and who received the viral inoculation.
Measure: Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
log10 copies/mL |  | 3.57 [2.67 to 4.46] |  |  | 3.37 [2.47 to 4.26]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other; p = 0.756, ANOVA; Difference in Least Squares Mean = 0.20, 95% CI 2-sided [-1.07 to 1.47]

28. Secondary Outcome: Part 2: Percentage of Participants With qRT-PCR-Confirmed Influenza Infection From Day 1 PM up to Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: The percentage of participants with two quantifiable (≥ LLOQ) influenza challenge virus qRT-PCR measurements reported on ≥2 independent nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening) within 48 hrs of each other, starting from baseline (Day 1 PM) up to planned discharge from quarantine (Day 8, AM). qRT-PCR-confirmed influenza infection in Part 2 participants from day 1 PM up to day 8 is presented. Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
Percentage of participants |  | 40.00 [23.87 to 57.89] |  |  | 40.00 [23.87 to 57.89]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other — Clopper and Pearson exact binomial method; Difference in Percentage = 0.00, 95% CI 2-sided [-23.21 to 23.21]

29. Secondary Outcome: Part 2: Percentage of Participants With qRT-PCR-Confirmed Symptomatic Influenza Infection From Day 1 PM up to Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: The percentage of participants with two quantifiable (≥ LLOQ) influenza challenge virus qRT-PCR measurements reported on ≥2 independent nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening) within 48 h of each other, starting from baseline (Day 1 PM) up to planned discharge from quarantine (Day 8, AM) AND total symptom score (TSS) ≥2 at ≥1 time point following inoculation. Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom is used to obtain TSS. Total symptom scores (TSS) ranged from 0 to 31, with higher scores indicating greater symptom severity. Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
Percentage of participants |  | 37.14 [21.47 to 55.08] |  |  | 40.00 [23.87 to 57.89]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other — Clopper and Pearson binomial method; Difference in percentage = -2.86, 95% CI 2-sided [-25.78 to 20.27]

30. Secondary Outcome: Part 2: Percentage of Participants With qRT-PCR-Confirmed Moderately Severe Symptomatic Influenza Infection From Day 1 PM up to Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: The percentage of participants with two quantifiable (≥ LLOQ) influenza challenge virus qRT-PCR measurements reported on ≥2 independent nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening) over 2 days AND any symptom of Grade ≥2 at ≥1 timepoint following inoculation. Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from Grade 0 ("no symptoms") to Grade 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from Grade 0 ("no symptoms") to Grade 4 ("symptoms at rest"). Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
Percentage of participants |  | 25.71 [12.49 to 43.26] |  |  | 34.29 [19.13 to 52.21]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other — Clopper and Pearson exact binomial method; Difference in Percentage = -8.57, 95% CI 2-sided [-30.26 to 13.38]

31. Secondary Outcome: Part 2: Percentage of Participants With qRT-PCR-Confirmed Febrile Influenza Infection From Day 1 PM up to Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: Percentage of participants with qRT-PCR-confirmed febrile influenza infection was defined as the percentage of participants with two quantifiable (≥ LLOQ) influenza challenge virus qRT-PCR measurements reported on ≥2 independent nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening) over 2 days, starting from baseline (Day 1 PM) up to planned discharge from quarantine (Day 8, am) AND a temperature of ≥37.9°C at ≥1 time point following inoculation. Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
Percentage of participants |  | 17.14 [6.56 to 33.65] |  |  | 22.86 [10.42 to 40.14]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other — Clopper and Pearson binomial method; Difference in percentage = -5.71, 95% CI 2-sided [-25.18 to 13.97]

32. Secondary Outcome: Part 2: Percentage of Participants With QVC Confirmed Influenza Infection From Day 1 PM up to Day 8 AM After Intranasal Inoculations (Molnupiravir PEP and Placebo)
Description: Percentage of participants with QVC confirmed influenza infection was defined as the percentage of participants with one quantifiable ≥LLOQ influenza challenge virus measurement from QVC (TCID50 assay) from a nasopharyngeal sample (nasal wash samples collected twice daily - morning and evening). Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
Percentage of Participants |  | 17.14 [6.56 to 33.65] |  |  | 22.86 [10.42 to 40.14]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other — Clopper and Pearson binomial method; Difference in percentage = -5.71, 95% CI 2-sided [-25.18 to 13.97]

33. Secondary Outcome: Part 2: Percentage of Participants With QVC Confirmed Symptomatic Influenza Infection From Day 1 PM up to Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: Percentage of participants with QVC (TCID50 assay) confirmed symptomatic influenza infection was defined as the percentage of participants with one quantifiable ≥LLOQ influenza challenge virus measurement from quantitative viral culture from a nasopharyngeal sample (nasal wash samples collected twice daily - morning and evening) AND TSS ≥2 at ≥1 time point following inoculation. Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom is used to obtain a total symptom score (TSS). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
Percentage of Participants |  | 14.29 [4.81 to 30.26] |  |  | 22.86 [10.42 to 40.14]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other — Clopper and Pearson binomial method; Difference in percentage = -8.57, 95% CI 2-sided [-27.63 to 10.50]

34. Secondary Outcome: Part 2: Duration of Quantifiable Infection Determined by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: Duration of quantifiable infection was defined as the time in days from the first quantifiable (≥LLOQ) influenza challenge virus measurement until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure (after which there are no more confirmed quantifiable samples) determined by qRT-PCR. Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 17 | 0 | 0 | 16
Days |  | 2.61 (1.87) |  |  | 3.03 (1.44)

35. Secondary Outcome: Part 2: Duration of Quantifiable Infection Determined by QVC From Day 1 PM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: Duration of quantifiable infection was defined as the time in days from the first quantifiable (≥LLOQ) influenza challenge virus measurement until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure after which there are no more confirmed quantifiable samples) determined by QVC (TCID50 assay). Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 6 | 0 | 0 | 8
Days |  | 0.58 (0.21) |  |  | 1.37 (0.68)

36. Secondary Outcome: Part 2: Time to Confirmed Negative Test Determined by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: Time to confirmed negative test was defined as the time in days from baseline until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure (after which there are no more confirmed quantifiable samples) as determined by qRT-PCR from nasal wash samples collected twice daily (morning and evening). Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
Days |  | 0.0 [0.0 to 3.0] |  |  | 0.0 [0.0 to 1.5]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other; p = 0.3102, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.51 to 1.33] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

37. Secondary Outcome: Part 2: Time to Confirmed Negative Test Determined by QVC (TCID50 Assay) From Day 1 PM Through Day 8 AM After Intranasal Inoculations (Molnupiravir PEP and Placebo)
Description: Time to confirmed negative test was defined as the time in days from baseline until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure (after which there are no more confirmed quantifiable samples) as determined by QVC (TCID50 assay) from nasal wash samples collected twice daily (morning and evening). Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
Days |  | 0.7 [0.0 to 1.5] |  |  | 0.0 [0.0 to 0.5]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other; p = 0.0779, Log Rank; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.27 to 1.14] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

38. Secondary Outcome: Part 2: Time to PVL Determined by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: Time to PVL was defined as the time in days from the baseline until the PVL measurement as determined by qRT-PCR from nasal wash samples collected twice daily (morning and evening). PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples. Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM Up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
Days |  | 0.66 (1.01) |  |  | 1.04 (1.58)

39. Secondary Outcome: Part 2: Time to PVL Determined by QVC From Day 1 PM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: Time to PVL was defined as the time in days from the baseline until the PVL measurement as determined by QVC (TCID50 assay) from nasal wash samples collected twice daily (morning and evening). PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples. Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 17 | 0 | 0 | 16
Days |  | 0.74 (0.79) |  |  | 1.47 (1.43)

40. Secondary Outcome: Part 2: VL-AUC Determined by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx and Placebo)
Description: VL-AUC is the area under the viral load-time curve of influenza challenge virus nasopharyngeal samples determined by qRT-PCR. H1N1 viral load was computed for each participant from nasophayngeal samples collected twice daily (morning and evening) from day 1 PM to day 8 AM. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for Molnupiravir Tx and placebo were presented for this endpoint.
Time Frame: Day 1 PM, Days 2, 3, 4, 5, 6, 7 - twice daily (AM and PM), and day 8 AM post viral inoculation
Population: All randomized participants who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, meet the criterion for laboratory-confirmed influenza infection and had available data for the endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: day*log10 copies/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 0 | 14
day*log10 copies/mL |  |  | 14.40 [11.75 to 17.06] |  | 18.19 [15.63 to 20.75]
Statistical Analysis 1: Comparison: Molnupiravir Treatment (Tx) vs Placebo; Test type: Other; p = 0.045, ANOVA; Difference in Least Squares Mean = -3.79, 95% CI 2-sided [-7.47 to -0.10]

41. Secondary Outcome: Part 2: VL-AUC Determined by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation (OTV Tx and Placebo)
Description: VL-AUC is the area under the viral load-time curve of influenza challenge virus nasopharyngeal samples determined by qRT-PCR. H1N1 viral load was computed for each participant from nasophayngeal samples collected twice daily (morning and evening) from day 1 PM to day 8 AM. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for OTV Tx and placebo were presented for this endpoint.
Time Frame: Day 1 PM, Days 2, 3, 4, 5, 6, 7 - twice daily (AM and PM), and day 8 AM post viral inoculation
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: day*log10 copies/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 15 | 14
day*log10 copies/mL |  |  |  | 15.62 [12.67 to 18.58] | 18.19 [15.13 to 21.24]
Statistical Analysis 1: Comparison: Oseltamivir (OTV) Tx vs Placebo; Test type: Other; p = 0.226, ANOVA; Difference in Least Squares Mean = -2.56, 95% CI 2-sided [-6.81 to 1.69]

42. Secondary Outcome: Part 2: VL-AUC Determined by Quantitative Viral Culture (TCID50 Assay) From Day 1 PM Through Discharge Day 8 AM After Intranasal Inoculation (Molnupiravir Tx and Placebo)
Description: VL-AUC is the area under the viral load-time curve of influenza challenge virus nasopharyngeal samples determined by QVC. H1N1 viral load was computed for each participant from nasophayngeal samples collected twice daily (morning and evening) from day 1 PM to day 8 AM. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for Molnupiravir Tx and placebo were presented for this endpoint.
Time Frame: Day 1 PM, Days 2, 3, 4, 5, 6, 7 - twice daily (AM and PM), and day 8 AM post viral inoculation
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: day*log10 TCID50/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 0 | 14
day*log10 TCID50/mL |  |  | 2.74 [1.40 to 4.09] |  | 4.34 [3.05 to 5.64]
Statistical Analysis 1: Comparison: Molnupiravir Treatment (Tx) vs Placebo; Test type: Other; p = 0.090, ANOVA; Difference in Least Squares Mean = -1.60, 95% CI 2-sided [-3.47 to 0.27]

43. Secondary Outcome: Part 2: VL-AUC Determined by Quantitative Viral Culture (TCID50 Assay) From Day 1 PM Through Day 8 AM After Intranasal Inoculation (OTV Tx and Placebo)
Description: VL-AUC is the area under the viral load-time curve of influenza challenge virus nasopharyngeal samples determined by QVC. H1N1 viral load was computed for each participant from nasopharyngeal samples collected twice daily (morning and evening) from day 1 PM to day 8 AM. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for OTV Tx and placebo were presented for this endpoint.
Time Frame: Day 1 PM, Days 2, 3, 4, 5, 6, 7 - twice daily (AM and PM), and day 8 AM post viral inoculation
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: day*log10 TCID50/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 15 | 14
day*log10 TCID50/mL |  |  |  | 5.08 [3.05 to 7.11] | 4.34 [2.24 to 6.45]
Statistical Analysis 1: Comparison: Oseltamivir (OTV) Tx vs Placebo; Test type: Other; p = 0.609, ANOVA; Difference in Least Squares Mean = 0.74, 95% CI 2-sided [-2.19 to 3.66]

44. Secondary Outcome: Part 2: PVL Determined by Quantitative Viral Culture (TCID50 Assay) From Day 1 PM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx and Placebo)
Description: PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening). PVL as determined by quantitative viral culture (QVC) was measured starting from day 1 PM (baseline) up to planned discharge from quarantine (day 8 AM). PVL of the H1N1 strain was measured by quantitative viral culture (QVC) using TCID50 assay and analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for Molnupiravir Tx and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 TCID 50/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 0 | 14
log10 TCID 50/mL |  |  | 3.33 [2.34 to 4.32] |  | 2.99 [2.03 to 3.95]
Statistical Analysis 1: Comparison: Molnupiravir Treatment (Tx) vs Placebo; Test type: Other — Difference in Least Squares Mean; p = 0.614, ANOVA; Difference in Least Squares Mean = 0.34, 95% CI 2-sided [-1.04 to 1.72]

45. Secondary Outcome: Part 2: PVL Determined by Quantitative Viral Culture (TCID50 Assay) From Day 1 PM Through Day 8 AM After Intranasal Inoculation (OTV Tx and Placebo)
Description: PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening). PVL as determined by quantitative viral culture (QVC) was measured starting from day 1 PM (baseline) up to planned discharge from quarantine (day 8 AM). PVL of the H1N1 strain was measured by quantitative viral culture (QVC) using TCID50 assay and analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for OTV Tx and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 TCID 50/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 15 | 14
log10 TCID 50/mL |  |  |  | 3.36 [2.34 to 4.37] | 2.99 [1.94 to 4.04]
Statistical Analysis 1: Comparison: Molnupiravir Treatment (Tx) vs Placebo; Test type: Other; p = 0.608, ANOVA; Difference in Least Squares Mean = 0.37, 95% CI 2-sided [-1.09 to 1.83]

46. Secondary Outcome: Part 2: PVL Determined by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx and Placebo)
Description: PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening) from day 1 PM (baseline) through day 8 AM. PVL of the H1N1 strain was measured by qRT-PCR and analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for Molnupiravir Tx and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 0 | 14
log10 copies/mL |  |  | 6.74 [6.15 to 7.33] |  | 6.31 [5.74 to 6.88]
Statistical Analysis 1: Comparison: Molnupiravir Treatment (Tx) vs Placebo; Test type: Other; p = 0.288, ANOVA; Difference in Least Squares Mean = 0.43, 95% CI 2-sided [-0.39 to 1.25]

47. Secondary Outcome: Part 2: PVL Determined by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation (OTV Tx and Placebo)
Description: PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening) from day 1 PM (baseline) through day 8 AM. PVL of the H1N1 strain was measured by qRT-PCR and analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for OTV Tx and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 15 | 14
log10 copies/mL |  |  |  | 6.39 [5.78 to 7.01] | 6.31 [5.67 to 6.94]
Statistical Analysis 1: Comparison: Oseltamivir (OTV) Tx vs Placebo; Test type: Other; p = 0.842, ANOVA; Difference in Least Squares Mean = 0.09, 95% CI 2-sided [-0.80 to 0.97]

48. Secondary Outcome: Part 2: Duration of Quantifiable Infection Determined by qRT-PCR From Day 2 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx, OTV Tx and Placebo)
Description: Duration of quantifiable infection was defined as the time from the first quantifiable (≥LLOQ) influenza challenge virus measurement until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure (after which there are no more confirmed quantifiable samples) determined by qRT-PCR. Per protocol, only data for Molnupiravir Tx, OTV Tx and placebo were presented for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 15 | 14
Days |  |  | 2.16 (0.95) | 2.67 (1.79) | 3.25 (0.89)

49. Secondary Outcome: Part 2: Duration of Quantifiable Infection Determined by QVC From Day 2 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx, OTV Tx and Placebo)
Description: Time from the first quantifiable (≥LLOQ) influenza challenge virus measurement until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure after which there are no more confirmed quantifiable samples) determined by QVC (TCID50 assay). Per protocol, only data for Molnupiravir Tx, OTV Tx and placebo were presented for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 9 | 10 | 8
Days |  |  | 0.85 (0.43) | 1.90 (1.31) | 1.19 (0.52)

50. Secondary Outcome: Part 2: Time to Confirmed Negative Test Determined by qRT-PCR From Day 2 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx and Placebo)
Description: Time to confirmed negative test was defined as the time in days from baseline until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure (after which there are no more confirmed quantifiable samples) as determined by qRT-PCR from nasal wash samples collected twice daily (morning and evening). Per protocol, only data for Molnupiravir Tx and placebo were presented for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 0 | 14
Days |  |  | 2.5 [1.5 to 2.5] |  | 3.7 [2.5 to 4.5]
Statistical Analysis 1: Comparison: Molnupiravir Treatment (Tx) vs Placebo; Test type: Other; p = 0.0042, Log Rank; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.14 to 0.71] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

51. Secondary Outcome: Part 2: Time to Confirmed Negative Test Determined by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation (OTV Tx and Placebo)
Description: Time to confirmed negative test was defined as the time in days from baseline until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure (after which there are no more confirmed quantifiable samples) as determined by qRT-PCR from nasal wash samples collected twice daily (morning and evening). Per protocol, only data for OTV Tx and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 15 | 14
Days |  |  |  | 2.0 [1.0 to 4.0] | 3.7 [2.5 to 4.5]
Statistical Analysis 1: Comparison: Molnupiravir Treatment (Tx) vs Placebo; Test type: Other; p = 0.3290, Log Rank; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.33 to 1.46] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

52. Secondary Outcome: Part 2: Time in Days to Confirmed Negative Test Determined by QVC From Day 2 AM Through Day 8 AM After Intranasal Inoculations (Molnupiravir Tx and Placebo)
Description: Time to confirmed negative test was defined as the time in days from baseline until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure (after which there are no more confirmed quantifiable samples) as determined by QVC (TCID50 assay) from nasal wash samples collected twice daily (morning and evening). Per protocol, only data for Molnupiravir Tx and placebo were presented for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 0 | 14
Days |  |  | 0.5 [0.0 to 1.0] |  | 1.0 [0.0 to 1.5]
Statistical Analysis 1: Comparison: Molnupiravir Treatment (Tx) vs Placebo; Test type: Other; p = 0.1502, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.27 to 1.34] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

53. Secondary Outcome: Part 2: Time in Days to Confirmed Negative Test Determined by QVC From Day 2 AM Through Day 8 AM After Intranasal Inoculation (OTV Tx and Placebo)
Description: Time to confirmed negative test was defined as the time from baseline until the first confirmed unquantifiable (<LLOQ detected or not detected) assessment after the peak measure (after which there are no more confirmed quantifiable samples) as determined by QVC (TCID50 assay) from nasal wash samples collected twice daily (morning and evening). Per protocol, only data for OTV Tx and placebo were presented for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 15 | 14
Days |  |  |  | 1.0 [0.0 to 1.5] | 1.0 [0.0 to 1.5]
Statistical Analysis 1: Comparison: Molnupiravir Treatment (Tx) vs Placebo; Test type: Other; p = 0.4865, Log Rank; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.59 to 2.92] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

54. Secondary Outcome: Part 2: Time to PVL Determined by qRT-PCR From Day 1 PM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx, OTV Tx and Placebo)
Description: Time to PVL was defined as the time in days from the baseline until the PVL measurement as determined by qRT-PCR from nasal wash samples collected twice daily (morning and evening). PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples. Per protocol, only data for Molnupiravir Tx, OTV Tx and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 15 | 14
Days |  |  | 0.19 (0.33) | 0.43 (0.26) | 1.53 (1.56)

55. Secondary Outcome: Part 2: Time to PVL Determined by QVC From Day 2 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx, OTV and Placebo)
Description: Time to PVL was defined as the time in days from the baseline until the PVL measurement as determined by QVC (TCID50 assay) from nasal wash samples collected twice daily (morning and evening). PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples. Per protocol, only data for Molnupiravir Tx, OTV Tx and placebo were presented for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 15 | 14
Days |  |  | 0.11 (0.22) | 0.37 (0.30) | 1.14 (1.45)

56. Secondary Outcome: Part 2: Total Symptom Score AUC (TSS-AUC) From Day 2 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom was used to obtain TSS. Total symptom scores (TSS) ranged from 0 to 31, with higher scores indicating greater symptom severity. TSS were used to calculate the AUC for each participant based on the available non-missing calculated total symptom scores between Day 2 until Day 8 (quarantine discharge) using the Trapezoidal rule. TSS-AUC measured from 10 symptoms assessed 3 times daily within the graded symptom scoring was reported. Per protocol, only Molnupiravir Tx and placebo were included in the model.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale*Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 0 | 14
Scores on a Scale*Days |  |  | 14.72 [7.83 to 21.61] |  | 19.51 [12.87 to 26.15]
Statistical Analysis 1: Comparison: Molnupiravir Treatment (Tx) vs Placebo; Test type: Other; p = 0.313, ANOVA; Difference in Least Squares Mean = -4.79, 95% CI 2-sided [-14.36 to 4.78]

57. Secondary Outcome: Part 2: Total Symptom Score AUC (TSS-AUC) From Day 2 AM Through Day 8 AM After Intranasal Inoculation (OTV Tx and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). Total symptom scores (TSS) ranged from 0 to 31, with higher scores indicating greater symptom severity. For each participant, the sum of grade values for each symptom was used to obtain a total symptom score (TSS). TSS were used to calculate the AUC for each participant based on the available non-missing calculated total symptom scores between Day 2 until Day 8 (quarantine discharge) using the Trapezoidal rule. TSS-AUC was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only OTV Tx and placebo were included in the model. TSS-AUC measured from 10 symptoms within the graded symptom scoring was reported.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale*Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 15 | 14
Scores on a Scale*Days |  |  |  | 12.64 [6.22 to 19.05] | 19.51 [12.87 to 26.15]
Statistical Analysis 1: Comparison: Oseltamivir (OTV) Tx vs Placebo; Test type: Other; p = 0.138, ANOVA; Difference in Least Squares Mean = -6.87, 95% CI 2-sided [-16.11 to 2.36]

58. Secondary Outcome: Part 2: Peak TSS From Day 2 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom was used to obtain TSS. TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. The highest TSS (defined as the sum of all 10 individual composite symptoms) was summarized by treatment group and analyzed using a linear model with treatment group as a fixed categorical effect. Peak TSS measured from 10 symptoms within the graded symptom scoring system collected 3 times daily was reported. Per protocol, only Molnupiravir Tx and placebo were reported for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: All randomized participants who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation and meet the criterion for laboratory-confirmed influenza infection and had available data for the endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 0 | 14
Scores on a Scale |  |  | 9.38 [6.50 to 12.27] |  | 8.64 [5.87 to 11.42]
Statistical Analysis 1: Comparison: Molnupiravir Treatment (Tx) vs Placebo; Test type: Other; p = 0.706, ANOVA; Difference in LS mean = 0.74, 95% CI 2-sided [-3.26 to 4.74]

59. Secondary Outcome: Part 2: Peak TSS From Day 2 AM Through Day 8 AM After Intranasal Inoculation (OTV Tx and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom was used to obtain TSS. TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. The highest TSS (defined as the sum of all 10 individual composite symptoms) was summarized by treatment group and analyzed using a linear model with treatment group as a fixed categorical effect. Peak TSS measured from 10 symptoms within the graded symptom scoring system collected 3 times daily was reported was reported. Per protocol, only OTV Tx and Placebo were reported for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 15 | 14
Scores on a Scale |  |  |  | 7.07 [4.62 to 9.51] | 8.64 [6.11 to 11.18]
Statistical Analysis 1: Comparison: Oseltamivir (OTV) Tx vs Placebo; Test type: Other; p = 0.367, ANOVA; Difference in LS mean = -1.58, 95% CI 2-sided [-5.10 to 1.95]

60. Secondary Outcome: Part 2: Daily Maximum TSS From Day 2 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx, OTV Tx and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. For each participant, the sum of grade values for each symptom was used to obtain TSS. Maximum TSS on each day, measured by graded symptom scoring system collected 3 times daily were reported. Per protocol, only Molnupiravir Tx, OTV Tx and Placebo were reported for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 15 | 14
Scores on a Scale
  Day 2 |  |  | 9.15 (4.72) | 6.93 (4.06) | 7.57 (5.79)
  Day 3 |  |  | 7.08 (4.07) | 5.27 (3.67) | 6.50 (5.32)
  Day 4 |  |  | 4.31 (3.01) | 3.40 (2.26) | 5.86 (4.20)
  Day 5 |  |  | 1.69 (1.32) | 2.27 (1.62) | 3.71 (2.92)
  Day 6 |  |  | 0.62 (0.65) | 0.80 (1.08) | 2.57 (2.65)
  Day 7 |  |  | 0.31 (0.48) | 0.47 (0.99) | 1.50 (2.35)
  Day 8 |  |  | 0.00 (0.00) | 0.07 (0.26) | 0.57 (1.22)

61. Secondary Outcome: Part 2: Daily Maximum TSS From Day 1 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. For each participant, the sum of grade values for each symptom was used to obtain TSS. Maximum TSS on each day, measured by graded symptom scoring system collected 3 times daily were reported. Per protocol, only Molnupiravir PEP and Placebo were included in the model.
Time Frame: From Day 1 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
Scores on a Scale
  Day 1 |  | 2.20 (3.08) |  |  | 1.94 (2.25)
  Day 2 |  | 4.09 (4.47) |  |  | 4.71 (5.06)
  Day 3 |  | 2.69 (2.59) |  |  | 4.09 (4.63)
  Day 4 |  | 1.80 (1.89) |  |  | 3.38 (3.80)
  Day 5 |  | 1.11 (1.69) |  |  | 2.06 (2.52)
  Day 6 |  | 0.71 (1.27) |  |  | 1.26 (2.14)
  Day 7 |  | 0.31 (0.63) |  |  | 0.82 (1.73)
  Day 8 |  | 0.26 (0.66) |  |  | 0.24 (0.82)

62. Secondary Outcome: Part 2: Duration of Grade ≥2 Symptoms From Day 2 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx, OTV Tx and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from Grade 0 ("no symptoms") to Grade 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from Grade 0 ("no symptoms") to Grade 4 ("symptoms at rest"). Duration in days of Grade ≥2 symptoms was defined as the duration of time in days from the first occurrence of any symptom assigned Grade 2 or higher, to the beginning of the first 24-hour period without any symptom assigned Grade 2 or higher, after the peak TSS. Per protocol, Molnupiravir Tx, OTV Tx and Placebo were included in the analysis.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 12 | 11 | 11
Days |  |  | 2.16 (1.12) | 2.10 (1.40) | 2.43 (1.32)

63. Secondary Outcome: Part 2: Time to Symptom Resolution From Day 2 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx, OTV Tx and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. Time in days to symptom resolution was defined as the time in days until the beginning of a 24-hour period with no symptoms above the baseline maximum TSS, as measured by graded symptom scoring system collected 3 times daily. Baseline maximum is defined as the maximum TSS on Day -1 (1 day prior to intranasal inoculation). Per protocol, only Molnupiravir Tx, OTV Tx and Placebo were presented for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: All randomized participants who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation and meet the criterion for laboratory-confirmed influenza infection.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 14 | 11
Days |  |  | 3.78 (1.33) | 3.48 (1.23) | 4.07 (1.50)

64. Secondary Outcome: Part 2: Time to Peak TSS From Day 2 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx, OTV Tx and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom was used to obtain TSS. TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. The highest total symptom score recorded on each day, across the three assessments, for each participant was summarized descriptively by treatment group and assessment day. Time to peak TSS was defined as the time from the assessment at Day 2 AM until the highest total symptom score was calculated. Per protocol, only Molnupiravir Tx, OTV Tx and Placebo were presented for this endpoint.
Time Frame: From Day 2 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 15 | 14
Days |  |  | 0.25 (0.40) | 0.14 (0.25) | 0.90 (1.12)

65. Secondary Outcome: Part 2: Total Symptom Score AUC (TSS-AUC) From Day 1 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom was used to obtain TSS. Total symptom scores (TSS) ranged from 0 to 31, with higher scores indicating greater symptom severity. TSS were used to calculate the AUC for each participant based on the available non-missing calculated total symptom scores between Day 1 until Day 8 (quarantine discharge) using the Trapezoidal rule. Per protocol, only Molnupiravir PEP and Placebo was included in the model.
Time Frame: From Day 1 AM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale*Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
Scores on a Scale*Days |  | 8.84 [4.55 to 13.12] |  |  | 12.98 [8.70 to 17.27]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other; p = 0.177, ANOVA; Difference in LS Mean = -4.14, 95% CI 2-sided [-10.20 to 1.92]

66. Secondary Outcome: Part 2: Peak TSS From Day 1 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom is used to obtain TSS. TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. The highest TSS (defined as the sum of all 10 individual composite symptoms) was summarized by treatment group and analyzed using a linear model with treatment group as a fixed categorical effect. Peak TSS measured from 10 symptoms within the graded symptom scoring system collected 3 times daily was reported. Per protocol, only Molnupiravir PEP and Placebo were presented for this endpoint.
Time Frame: From Day 1 AM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 0 | 0 | 35
Scores on a Scale |  | 4.66 [3.06 to 6.26] |  |  | 5.63 [4.03 to 7.23]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other; p = 0.395, ANOVA; Difference in LS mean = -0.97, 95% CI 2-sided [-3.24 to 1.29]

67. Secondary Outcome: Part 2: Duration of Grade ≥2 Symptoms From Day 1 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from Grade 0 ("no symptoms") to Grade 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from Grade 0 ("no symptoms") to Grade 4 ("symptoms at rest"). Duration of Grade 2 symptoms is defined as the duration in days from the first occurrence of a Grade 2 or higher symptom until the first 24 hours period where no Grade 2 or higher symptoms are recorded. Per protocol, Molnupiravir PEP and Placebo were included in the analysis.
Time Frame: From Day 1 AM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 13 | 0 | 0 | 19
Days |  | 1.78 (1.59) |  |  | 2.04 (1.43)

68. Secondary Outcome: Part 2: Time to Symptom Resolution From Day 1 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. Time in days to symptom resolution was defined as the time in days from the beginning of the specified time frame until the beginning of a 24-hour period with no symptoms above the baseline maximum TSS, as measured by graded symptom scoring system collected 3 times daily. Baseline maximum is defined as the maximum TSS on Day -1 (1 day prior to intranasal inoculation). Per protocol, only Molnupiravir PEP and Placebo are reported.
Time Frame: From Day 1 AM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 32 | 0 | 0 | 31
Days |  | 3.14 (2.16) |  |  | 3.44 (2.40)

69. Secondary Outcome: Part 2: Time to Peak TSS From Day 1 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). For each participant, the sum of grade values for each symptom is used to obtain TSS. TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. Time in days to peak TSS was defined as the time from baseline to the time of peak TSS measured by the graded symptom scoring system collected 3 times daily. Per protocol, only Molnupiravir PEP and Placebo are reported.
Time Frame: From Day 1 AM up to Day 8 post viral inoculation
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 28 | 0 | 0 | 31
Days |  | 1.77 (1.04) |  |  | 1.54 (1.21)

70. Secondary Outcome: Part 2: Number of Participants With One or More AE (Molnupiravir Tx and Molnupiravir PEP)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants with one or more AEs are presented. Per protocol, only Molnupiravir PEP and Molnupiravir Tx are reported.
Time Frame: Up to approximately 31 days
Population: All participants who received at least one dose of treatment in Molnupiravir PEP and Molnupiravir Tx groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 36 | 0 | 0
Participants |  | 8 | 11 |  |

71. Secondary Outcome: Part 2: Number of Participants Discontinuing Study Treatment Due to an AE (Molnupiravir Tx and Molnupiravir PEP)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinued study treatment due to an AE are presented. Per protocol, only Molnupiravir PEP and Molnupiravir Tx are reported.
Time Frame: Up to day 6
Population: All participants who received at least one dose of treatment in Molnupiravir PEP and Molnupiravir Tx groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 36 | 0 | 0
Participants |  | 0 | 0 |  |

72. Secondary Outcome: Number of Participants With One or More Viral Challenge-Related AE
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE is viral challenge-related as determined by investigator. The number of participants with one or more viral challenge-related AEs are presented.
Time Frame: Up to approximately 31 days
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 35 | 36 | 35 | 35
Participants | 9 | 1 | 2 | 3 | 6

73. Secondary Outcome: Part 2: Number of Participants With Concomitant Medication Use From Viral Challenge Through Day 28
Description: Concomitant medications were defined as any prescription medications, over the counter drugs or dietary supplements that a participant happened to be taking while on study, in addition to molnupiravir. The number of participants who use at least 1 concomitant medication from viral challenge (Day 0) through Day 28 were reported. Per protocol, only Molnupiravir PEP, Molnupiravir Tx, OTV Tx and Placebo were reported.
Time Frame: From Day 0 up to Day 28
Population: All participants who received at least one dose of treatment and used at least 1 concomitant medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 36 | 35 | 35
Participants |  | 18 | 10 | 10 | 17

74. Secondary Outcome: Maximum Plasma Concentration (Cmax) of N-hydroxycytidine (NHC)
Description: NHC is the pharmacologically active moiety of molnupiravir (MK-4482) and therefore its primary pharmacokinetic measure. Cmax was defined as the peak concentration of NHC over the dosing interval. Plasma samples were collected at multiple time points pre-and post-administration and used to determine Cmax following oral administration of Molnupiravir. Per protocol, Cmax for only Molnupiravir PEP and Molnupiravir Tx were reported.
Time Frame: Day (D) 0, D2, D4: predose D5: predose, 0.5, 1.5, 4, 8, 12, 24, 48, 72 hours post dose
Population: All participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model and had available data from at least one treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 36 | 0 | 0
ng/mL |  | 3730 (46.5) | 3680 (48.4) |  |

75. Primary Outcome: Part 1: Infectivity Rate Based on Quantitative Reverse Transcriptase-Polymerase Chain Reaction (qRT-PCR) From Day 1 PM Through Day 8 AM
Description: Infectivity rate was defined as the number of participants with two quantifiable (≥lower limit of quantitation (LLOQ)) influenza challenge virus (A/France/759/21 [H1N1] strain) qRT-PCR measurements reported on ≥2 independent nasopharyngeal samples (from nasal wash samples collected twice daily - morning and evening). Infectivity rate based on qRT-PCR in Part 1 participants from baseline (day 1 PM - afternoon) up to planned discharge from quarantine (day 8 AM - post viral inoculation) is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
Participants | 15 |  |  |  |

76. Primary Outcome: Part 1: Infectivity Rate Based on Quantitative Reverse Transcriptase-Polymerase Chain Reaction (qRT-PCR) From Day 2 PM Through Day 8 AM
Description: The number of participants with two quantifiable (≥lower limit of quantitation (LLOQ)) influenza challenge virus qRT-PCR measurements reported on ≥2 independent nasopharyngeal samples (from nasal wash samples collected twice daily - morning and evening). Infectivity rate based on qRT-PCR in Part 1 participants from day 2 PM up to day 8 post viral inoculation is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: From Day 2 PM up to Day 8 post viral inoculation
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
Participants | 14 |  |  |  |

77. Primary Outcome: Part 1: Number of Participants Experiencing ≥1 Viral Challenge-related Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE is viral challenge-related as determined by the investigator. Number of participants experiencing ≥1 viral challenge-related AE in part 1 is presented. Per protocol, only data for part 1 participants were presented for this endpoint.
Time Frame: Up to approximately 31 days
Population: All Part 1 participants who received viral inoculation and had available data for the endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 20 | 0 | 0 | 0 | 0
Participants | 9 |  |  |  |

78. Primary Outcome: Part 2: Peak Viral Load (PVL) Determined by Quantitative Viral Culture Tissue Culture Infective Dose 50% (TCID50) Assay From Day 1 PM Through Day 8 AM After Intranasal Inoculation (Molnupiravir PEP and Placebo)
Description: PVL was defined as the maximum viral load of influenza challenge virus from nasopharyngeal samples (nasal wash samples collected twice daily - morning and evening). PVL as determined by quantitative viral culture (QVC) was measured starting from day 1 PM (baseline) up to planned discharge from quarantine (day 8 AM). PVL of the H1N1 strain was measured by quantitative viral culture (QVC) using TCID50 plaque assay and analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for Molnupiravir PEP and placebo were presented for this endpoint.
Time Frame: From Day 1 PM up to Day 8 post viral inoculation
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 TCID50/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 17 | 0 | 0 | 16
log10 TCID50/mL |  | 1.85 [1.04 to 2.66] |  |  | 2.79 [1.96 to 3.62]
Statistical Analysis 1: Comparison: Molnupiravir Post-Exposure Prophylaxis (PEP) vs Placebo; Test type: Other — Difference in least squares mean; p = 0.110, ANOVA; Difference in least squares means = -0.94, 95% CI 2-sided [-2.10 to 0.22]

79. Primary Outcome: Part 2: Area Under the Viral Load-Time Curve (VL-AUC) Determined by QVC (TCID50 Assay) From Day 2 AM Through Day 8 AM After Intranasal Inoculation (Molnupiravir Tx and Placebo)
Description: VL-AUC is the area under the viral load-time curve of influenza challenge virus nasopharyngeal samples determined by QVC. H1N1 viral load was computed for each participant from nasopharyngeal samples collected twice daily (morning and evening) from day 2 AM to day 8 AM. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only data for Molnupiravir Tx and placebo were presented for this endpoint.
Time Frame: Days 2, 3, 4, 5, 6, 7 - twice daily (AM and PM), and day 8 AM post viral inoculation
Population: All randomized participants who received the viral inoculation, are influenza infected, have received at least 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into and had available data for the endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: day*log10 TCID50/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 0 | 13 | 0 | 14
day*log10 TCID50/mL |  |  | 2.74 [1.40 to 4.09] |  | 4.34 [3.05 to 5.64]
Statistical Analysis 1: Comparison: Molnupiravir Treatment (Tx) vs Placebo; Test type: Other; p = 0.090, ANOVA; Difference in least squares mean = -1.60, 95% CI 2-sided [-3.47 to 0.27]

80. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of NHC
Description: NHC is the pharmacologically active moiety of molnupiravir (MK-4482) and therefore its primary pharmacokinetic measure. Tmax was defined as the time to peak concentration. Plasma samples were collected at multiple time points pre-and post-administration and used to determine Tmax following oral administration of Molnupiravir. Per protocol, Tmax for only Molnupiravir PEP and Molnupiravir Tx were reported.
Time Frame: Day (D) 0, D2, D4: predose D5: predose, 0.5, 1.5, 4, 8, 12, 24, 48, 72 hours post dose
Population: as for outcome 74
Measure: Median (Full Range); unit: hr
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 36 | 0 | 0
hr |  | 1.68 [1.5 to 4.18] | 1.69 [1.47 to 4.38] |  |

81. Secondary Outcome: Area Under the Plasma Concentration From 0 to 12 Hours Postdose (AUC0-12) of NHC
Description: NHC is the pharmacologically active moiety of molnupiravir (MK-4482) and therefore its primary pharmacokinetic measure. Plasma samples were collected at multiple time points pre-and post-administration and used to determine the area under the plasma concentration curve from time 0 to 12 hours (AUC0-12) following oral administration of Molnupiravir. Per protocol, AUC0-12 for only Molnupiravir PEP and Molnupiravir Tx were reported.
Time Frame: Day (D) 0, D2, D4: predose D5: predose, 0.5, 1.5, 4, 8, 12 hours post dose
Population: as for outcome 74
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 36 | 0 | 0
hr*ng/mL |  | 9870 (28.5) | 9460 (27.7) |  |

82. Secondary Outcome: Area Under the Plasma Concentration From Dosing to Last Measurable Concentration (AUC0-Last) of NHC
Description: NHC is the pharmacologically active moiety of molnupiravir (MK-4482) and therefore its primary pharmacokinetic measure. AUC0-last is a measure of total exposure to Molnupiravir in plasma from the start of dosing to the time of the last quantifiable (<LLOQ]) sample. Per protocol, AUC0-Last for only Molnupiravir PEP and Molnupiravir Tx were reported.
Time Frame: Day (D) 0, D2, D4: predose D5: predose, 0.5, 1.5, 4, 8, 12, 24, 48, 72 hours post dose
Population: as for outcome 74
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 36 | 0 | 0
hr*ng/mL |  | 10300 (28.1) | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to too few pharmacokinetic (PK) sampling timepoints. |  |

83. Secondary Outcome: Ctrough of NHC
Description: NHC is the pharmacologically active moiety of molnupiravir (MK-4482) and therefore its primary pharmacokinetic measure. The trough concentration (Ctrough) was defined as the lowest concentration before the next dose. Plasma samples were collected at multiple time points pre-and post-administration and used to determine Ctrough. Per protocol, Ctrough for only Molnupiravir PEP and Molnupiravir Tx were reported.
Time Frame: Day (D) 0, D2, D4: predose D5: predose, 0.5, 1.5, 4, 8, 12, 24, 48, 72 hours post dose
Population: as for outcome 74
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 35 | 36 | 0 | 0
ng/mL |  | 23.8 (45.6) | 21 (46.4) |  |

84. Secondary Outcome: t1/2 of NHC
Description: NHC is the pharmacologically active moiety of molnupiravir (MK-4482) and therefore its primary pharmacokinetic measure. t1/2 is the amount of time required to clear 50% of NHC following the oral administration of Molnupiravir. Per protocol, t1/2 for only Molnupiravir PEP and Molnupiravir Tx were reported.
Time Frame: Day (D) 0, D2, D4: predose D5: predose, 0.5, 1.5, 4, 8, 12, 24, 48, 72 hours post dose
Population: as for outcome 74
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
Number analyzed (Participants) | 0 | 34 | 36 | 0 | 0
hr |  | 22.1 (16.2) | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to too few pharmacokinetic (PK) sampling timepoints. |  |

ADVERSE EVENTS:
Time Frame: Up to approximately 31 days
Description: Analysis population for all-cause mortality consists of all allocated and randomized participants. Analysis population for safety consists of all participants who received viral inoculation or at least one dose of study intervention.
Arm/Group | Viral Inoculation (Part 1) | Molnupiravir Post-Exposure Prophylaxis (PEP) | Molnupiravir Treatment (Tx) | Oseltamivir (OTV) Tx | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/35 | 0/36 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/35 | 0/36 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 10/20 | 5/35 | 6/36 | 8/35 | 8/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viral Inoculation (Part 1) (N=20) | Molnupiravir Post-Exposure Prophylaxis (PEP) (N=35) | Molnupiravir Treatment (Tx) (N=36) | Oseltamivir (OTV) Tx (N=35) | Placebo (N=35)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 7 (7) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Authorship will be determined by mutual agreement and in line with ICMJE authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT05818124/Prot_SAP_000.pdf